CLINICAL TRIAL: NCT05121519
Title: A Randomized Controlled Trial to Assess Abstinence of Coffee Compared to Continued Consumption on Recurrent Atrial Fibrillation Following Cardioversion
Brief Title: Does Eliminating Coffee Avoid Fibrillation?
Acronym: DECAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-35115
Record Dates: First submitted 2021-10-26; First posted 2021-11-16 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation; Coffee
Keywords: atrial fibrillation; coffee; afib
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avoid (Experimental): Patients will undergo this intervention for up to 6 months, or whenever their AF or atrial flutter returns, whichever comes first.
  Interventions: Other: Avoid coffee
- Consume (Experimental): Patients will undergo this intervention for up to 6 months, or whenever their AF or atrial flutter returns, whichever comes first.
  Interventions: Other: Consume coffee

INTERVENTIONS:
Other: Consume coffee — Drink coffee regularly (recommend at least 1 cup of caffeinated coffee or one shot of espresso per day)
  Arms: Consume
Other: Avoid coffee — Abstain from coffee and other caffeinated products
  Arms: Avoid

SUMMARY:
Given both the increasing population impact of atrial fibrillation (AF) and the widespread consumption of coffee in society, determining an associated benefit or risk of coffee consumption on AF is of great clinical relevance. This study will evaluate the effect of randomly assigning participants undergoing cardioversion to coffee abstinence or coffee continuation over a 6 month period. This study will provide the first, randomized evaluation of coffee on AF outcomes and will provide important information on whether or not coffee has any effect on AF recurrence.

DETAILED DESCRIPTION:
The purpose of this study is to assess how abstinence of coffee compared to continued consumption affects recurrent atrial fibrillation (AF) following cardioversion. As one of the most consumed beverages in the world, whether coffee has any effect on health outcomes is of considerable interest to physicians, scientists, and individual consumers. While significant data exist on the potential impact of coffee on many cardiometabolic parameters, there is conflicting data on any role of coffee on AF.

Most studies so far have been observational in nature, limiting how much insight there is on the role of coffee on AF. This study proposes to directly compare AF outcomes for patients with AF that abstain from coffee versus those that continue coffee consumption.

A total of 200 AF patients undergoing cardioversion will be enrolled in this study (100 per arm), and followed for up to 6 months post cardioversion. Differences in AF recurrence and symptoms will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 21 years of age
* Sustained AF or atrial flutter (provided patient has a history of AF)
* Planned/scheduled direct current electrical cardioversion
* Consumption greater than or equal to one cup of coffee per day sometime in the past 5 years
* Willing and able to comply with coffee abstinence or continuation for at least 6 months
* Life expectancy of at least 6 months
* Willing and able to return and comply with scheduled phone follow up visits
* Willing and able to provide written informed consent

Exclusion Criteria:

* Established allergy or adverse reaction to coffee
* Stated inability to comply with coffee abstinence or continuation
* AF ablation in preceding 3 months or planned in next 3 months
* Recent cardiothoracic surgery in preceding 3 months
* Pregnancy or desire to get pregnant within next 6 months.
* Current enrollment in an investigation or study of a cardiovascular device or investigational drug that would interfere with this study
* Any other criteria, which would make the patient unsuitable to participate in this study as determined by the Principal Investigator (e.g., an uncontrolled drug and/or alcohol addiction)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with first confirmed clinical recurrence of AF or atrial flutter, or device-detected recurrence lasting longer than 30 seconds, analyzed as a time-to-event outcome | 6 months
  The number and rate of AF or atrial flutter recurrence following cardioversion in the coffee abstinence group and the continued coffee group will be compared

SECONDARY OUTCOMES:
Adverse events | 6 months
  Any change in the number and rate of adverse events before censorship, including myocardial infarction, stroke or transient ischaemic attack, heart failure exacerbation, syncope, emergency department visit, hospitalization, and death, will be compared
Recurrent atrial flutter or AF separately | 6 months
  Any change in the number and rate of recurrent atrial flutter or AF separately as incident outcomes will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Marcus, MD, MAS, Principal Investigator — University of California, San Francisco; Christopher X Wong, MBBS, PhD, Principal Investigator — University of Adelaide; Christopher C Cheung, MD, MPH, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (3):
- UCSF Parnassus, San Francisco, California, United States
- Royal Adelaide Hospital, Adelaide, Australia
- Sunnybrook Health Science Centre, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong CX, Cheung CC, Montenegro G, Oo HH, Pena IJ, Tang JJ, Tu SJ, Wall G, Dewland TA, Moss JD, Gerstenfeld EP, Tseng ZH, Hsia HH, Lee RJ, Olgin JE, Vedantham V, Scheinman MM, Lee C, Sanders P, Marcus GM. Caffeinated Coffee Consumption or Abstinence to Reduce Atrial Fibrillation: The DECAF Randomized Clinical Trial. JAMA. 2026 Jan 27;335(4):317-325. doi: 10.1001/jama.2025.21056. PMID 41206802

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT05121519/Prot_SAP_006.pdf
  • Informed Consent Form (2024-08-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT05121519/ICF_007.pdf